CLINICAL TRIAL: NCT03055962
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study to Evaluate the Safety and Tolerability of a Once Daily Dose of 50 mg E2609 in Healthy Japanese Subjects
Brief Title: Study to Evaluate the Safety and Tolerability of a Once Daily Dose of 50 mg E2609 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: E2609-J081-014
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; E2609; Pharmacokinetics; Japan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E2609 50 mg (Experimental): Participants will receive E2609 50 milligrams (mg) orally once a day for 14 days.
  Interventions: Drug: E2609
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2609 — tablet
  Arms: E2609 50 mg
Drug: Placebo — tablet
  Arms: Placebo

SUMMARY:
Study E2609-J081-014 is a single-center, randomized, double-blind, placebo-controlled study conducted to evaluate the safety and tolerability of multiple oral doses of E2609 50 milligrams (mg), administered once daily for 14 days, in healthy Japanese participants aged 50 to 85 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged 50 to 85 years, inclusive at time of consent
* Body mass index (BMI) of 17.6 to 32 kilograms per meters squared (kg/m^2) at Screening

Exclusion Criteria:

* Personal or family history of seizure disorder, symptomatic seizures (not including a history of simple febrile seizures in childhood) or any past or present medical condition which, in the opinion of the investigator has the potential to reduce seizure threshold (eg, history of head trauma or concussion, previous alcohol abuse, substance abuse)
* A history of cerebrovascular accident or non-vasovagal-related loss of consciousness
* Any clinically significant findings on neurological examination
* A family history of Long QT Syndrome or a presence of other risk factors for Torsades de Pointes (TDP), such as hypokalemia, hypomagnesemia, or hypocalcemia
* History of cardiac arrhythmias, ischemic heart disease, or cerebrovascular disease
* A history of gastrointestinal surgery that may affect the pharmacokinetic profile of E2609 (eg, hepatectomy, nephrotomy, digestive organ resection)
* A known history of clinically significant drug or food allergies or presently experiencing significant seasonal allergy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with any serious adverse event and number of participants with any non-serious adverse event | up to Day 35 (Termination/Visit 5)
  An adverse event is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A serious adverse event is defined as any adverse event occurring at any dose that results in any of the following outcomes: results in death; is life threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life function; results in a congenital anomaly/birth defect; or can be defined as any other important medical event.
Number of participants with an abnormal, clinically significant laboratory test value | Screening; Baseline; Days 4, 8, 11, 14, 20 (Out-Patient Follow-up), and 35 (Termination/Visit 5); up to Day 62 (unscheduled Follow-up visits)
  Laboratory test values will be assigned a low/normal/high (LNH) classification according to whether the value was below (L), within (N), or above (H) the laboratory parameter's reference range. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant vital sign value | Screening; Baseline; up to Day 62
  Vital sign measurements (ie, systolic and diastolic blood pressure [BP] [millimeters of mercury (mmHg)], heart rate [beats per minute], respiratory rate [breaths per minute], body temperature [centigrade]) will be obtained in the supine position by a validated method. Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant electrocardiogram (ECG) finding | Screening; Baseline; up to Day 62
  Twelve-lead standard ECGs will be recorded in triplicate. ECGs will be recorded after the participant has been in the supine position for at least 10 minutes before and during the reading. In addition, all ECGs will be obtained before blood draws. Clinical significance will be determined by the Investigator.
Clinical assessment of suicidality per the suicidality rating scale | Baseline (Day -1), 24 hours after dosing (Day 2), Day 15, Day 20, Day 35 (Termination/Visit 5), up to Day 62 (unscheduled Follow-up visits)
  The suicidality rating scale will rate a participant's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The decision to classify an isolated suicidality rating scale response as an adverse event will be exercised through medical and scientific judgment.
Mean quality of sleep score per the Waketime Questionnaire, if necessary | up to Day 62
  Participants reporting adverse events (AEs) relating to abnormal dreams, nightmares, or sleep terrors will be questioned using the Waketime Questionnaire which is comprised of 5 individual questions. A participant is asked to rate the quality of their sleep as: 1, Very sound or restful; 2, Sound or restful; 3, Average quality; 4, Restless; or 5, Very restless.

SECONDARY OUTCOMES:
Mean maximum observed concentration (Cmax) of E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: predose; 1, 2, 3, 4, 6, and 10 hours postdose
  Cmax is defined as the maximum observed concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered. Using non-compartmental analysis, plasma concentrations of E2609 and metabolites will be analyzed to determine Cmax. Cmax will be summarized as the mean and standard deviation for all participants.
Mean minimum observed concentration (Cmin) of E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: predose; 1, 2, 3, 4, 6, and 10 hours postdose
  Cmin is defined as the minimum observed concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered. Using non-compartmental analysis, plasma concentrations of E2609 and metabolites will be analyzed to determine Cmin. Cmin will be summarized as the mean and standard deviation for all participants.
Median time from dosing to reach Cmax (tmax) of E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: predose; 1, 2, 3, 4, 6, and 10 hours postdose
  Tmax is defined as the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered. Using non-compartmental analysis, plasma concentrations of E2609 and metabolites will be analyzed to determine Tmax. Tmax will be summarized as the median for all participants.
Mean area under the concentration-time curve (AUC) from time 0 to 24 hours for E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: 1, 2, 3, 4, 6, 10, and 24 hours postdose
  AUC represents the total drug exposure over a defined period of time. Plasma concentrations of E2609 and its metabolites will be analyzed using a non-compartmental analysis approach to determine individual participant estimates of AUC(0-24h). AUC(0-24h) will be summarized as the mean and standard deviation for all participants and will be expressed in nanograms x hour per milliliter (ng*hr/mL).
Mean terminal elimination half-life (t1/2) following the last day of dosing (Day 14) of E2609 and metabolites | Day 14: 1, 2, 3, 4, 6, 10, 24, 48, 72, 96, and 144 hours postdose
  Terminal half-life is the time it takes for a substance to lose half of its pharmacologic, physiologic, or radiologic activity. Plasma concentrations of E2609 and its metabolites will be analyzed using a non-compartmental analysis approach to determine t1/2. t1/2 will be summarized as the mean and standard deviation for all participants and will be expressed in hours.
Mean average concentration calculated as AUCss/tau (Css,av), where tau is the dosing interval, of E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: 1, 2, 3, 4, 6, 10, and 24 hours postdose
  Css,av is the average steady-state concentration of a drug. Steady state will be achieved when the rate of E2609 administration and the rate of E2609 elimination are equal. Plasma concentrations of E2609 and its metabolites will be analyzed using a non-compartmental analysis approach to determine the Css,av.
Mean accumulation ratio for AUC, Cmax, and Cmin (Rac) for E2609 and metabolites on Day 1 and Day 14 | Days 1 and 14: 1, 2, 3, 4, 6, 10, and 24 hours postdose
  Rac is equal to the ratio of the AUC during a dosage interval at steady state to the AUC of a dosage interval after the first dose. Plasma concentrations of E2609 and its metabolites will be analyzed using a non-compartmental analysis approach to determine Rac. Rac will be summarized as the mean and standard deviation for all participants
Apparent clearance at steady state (CLss/F) of E2609 on Day 14 | Day 14: 1, 2, 3, 4, 6, 10, 24, 48, 72, 96, and 144 hours postdose
  CLss/F is the rate and extent of absorption and clearance of E2609 from the plasma. Plasma concentrations of E2609 and metabolites will be analyzed using a non-compartmental analysis approach to determine CLss/F.
Number of participants with polymorphisms of N-acetyltransferase 2 (NAT2) | Day 1
  NAT2 genotyping will be conducted, and the predicted phenotype (eg, slow, intermediate, or rapid acetylators) will be used in the statistical analysis to evaluate the relative impact of NAT2 polymorphisms on plasma concentrations of E2609 and/or its metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site, Fukuoka, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No